CLINICAL TRIAL: NCT06315023
Title: Prospective, Single Arm, Registry-based Study to Evaluate the Real-world Use of the DETOUR™ System in US Patients
Brief Title: The Percutaneous Transmural Arterial Bypass -1 Study (Post Approval Registry)
Acronym: PTAB1
Status: Recruiting | Type: Observational
Sponsor: Endologix (Industry)
Collaborators: Fivos (Unknown); Massachusetts General Hospital (Other); Society for Vascular Surgery Patient Safety Organization (Other)
Responsible Party: Sponsor
Other Study IDs: CP-0029
Record Dates: First submitted 2024-03-11; First posted 2024-03-18 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Peripheral Arterial Disease; Symptomatic Femoropopliteal Lesions
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- As Treated: All patients that have received the therapy; patients treated within and outside the IFU criteria subgroups; male and female subgroups; and duplex imaging subgroups for arterial and venous observations.
  Interventions: Device: DETOUR System
- Imaging Cohort: Sites that are performing (arterial and venous) duplex ultrasound assessments according to the institution's standard practice will be asked to participate in the DUS imaging cohort. The Imaging sub-study will consist of 55 female and 55 male subjects from these sites. Duplex imaging at 1-, 12-, 24-, and 36-months post-procedure will be collected to assess the endpoints of graft patency and venous thrombus within the vein containing the graft (n=110).
  Interventions: Device: DETOUR System

INTERVENTIONS:
Device: DETOUR System — Percutaneous Transmural Arterial Bypass Therapy using the DETOUR™ System

SUMMARY:
The purpose of this post-market surveillance study will be to evaluate the real-world use of the DETOUR System in treated patients with symptomatic femoropopliteal lesions from 200 mm to 460 mm in length with chronic total occlusions (100 mm to 425 mm) or diffuse stenosis > 70% who may be considered suboptimal candidates for surgical or alternative endovascular treatments.

DETAILED DESCRIPTION:
A maximum of 450 subjects will be enrolled with a target study population of at least 200 evaluable female and 200 evaluable male participants at the 12-month post-procedure follow-up visit. A maximum of 200 US sites. Sites will be selected that participate or will participate in the VQI PVI Registry. Follow up visits/assessments will be completed at 1, 12, 24-, 36-, 48-, and 60-months post-procedure. Study enrollment is expected to conclude over 4 years. Follow up data at 1 year is expected to conclude in 5 years from enrollment, with 5-year follow up expected to conclude in 9 years from enrollment.

ELIGIBILITY:
Inclusion Criteria: Participants should be a candidate for the DETOUR System as assessed by the treating physician after review of the clinical and anatomic Indications for Use.

-

Exclusion Criteria: There are no exclusion criteria. All cases entered in the registry at participating institutions will be included up through the targeted goals per the enrollment plan.

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with symptomatic femoropopliteal lesions from 200 mm to 460 mm in length with chronic total occlusions (100 mm to 425 mm) or diffuse stenosis > 70% who may be considered suboptimal candidates for surgical or alternative endovascular treatments.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2023-10-06 (Actual); Primary Completion 2028-06-07 (Estimated); Study Completion 2032-06-07 (Estimated)

PRIMARY OUTCOMES:
Freedom from CD-TLR | 1 Year
  Primary Effectiveness outcome is patency as defined as Freedom from Clinical Driven Target Lesion Revascularization (CD-TLR)
Freedom from MAE | 30 Days
  Primary Safety outcome is freedom from a major adverse event (MAE) at 30 days post-procedure defined as any occurrence of the following events: Death, Clinically-Driven Target Lesion Revascularization (CD-TLR), and/or Major Amputation of the Treated Limb.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Salinas Valley Memorial Hospital, Salinas, California
  - University of Connecticut, Storrs, Connecticut
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - Delray Medical Center, Delray Beach, Florida
  - Beth Isreal Deaconess Medical Center, Boston, Massachusetts
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - NYU Langone Medical Center, New York, New York
  - Cleveland Clinic Main Campus, Cleveland, Ohio
  - University of Pennsylvania, West Chester, Pennsylvania
  - Main Line Health, Wynnewood, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided